CLINICAL TRIAL: NCT07311941
Title: Rapid Escalation of LipiD Lowering Therapy to Reduce RecUrrent Cardiovascular Event (REDUCE) : All Comers Study
Brief Title: Rapid Escalation of LipiD Lowering Therapy to Reduce RecUrrent Cardiovascular Event
Acronym: REDUCE-Lipid
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, GuangMing Tan, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2024.356
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hyperlipidemia; Cardio Vascular Disease
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Coronary Syndrome: Patient with acute coronary syndrome due to atherosclerotic coronary artery disease
- Chronic coronary syndrome: Patient with chronic coronary syndrome due to atherosclerotic coronary artery disease

SUMMARY:
Hyperlipidaemia especially elevation of low-density lipoprotein cholesterol (LDL-C) is known to be the main contributor to the development of atherosclerotic cardiovascular disease (ASCVD).

Lowering LDL-C have been shown to reduce the risk of ASCVD2,3. Both the American Heart Association (AHA) and the European Society of Cardiology (ESC) advocated aggressive LDL-C target with statin being the first-line lipid-lowering therapy (LLT). However, a significant portion of patients did not attain their LDL-C goal in our locality. Statin no adherence, low uptake of adjuvant non-statin LLT, and therapeutic inertia are few potential causes for not achieving the LDL-C target. ESC recommends repeating blood test in 6-8 weeks after addition or alternation of LLT, but this recommendation was not routinely followed in current local practice due to resources constrain.

This registry therefore aims to investigate the strategy of frequent monitoring of LDL-C and titration of LLT in achieving LDL-C treatment target at a dedicated specialist clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* (Cohort 1) Diagnosis of acute coronary syndrome due to atherosclerotic coronary artery disease
* (Cohort 2) Diagnosis of chronic coronary syndrome due to atherosclerotic coronary artery disease

Exclusion Criteria:

* Inability to provide valid consent by the patient or his legal guardian
* Diagnosis of ACS due to other causes than atherosclerotic coronary artery disease.
* Psychiatric or severe neurological disorder, cirrhosis, or active malignancy leading to a life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged greater than 18 and who are admitted for a diagnosis of acute coronary syndrome (ACS) due to atherosclerotic coronary artery disease based on invasive coronary angiography will be recruited into this registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol (LDL-C) level | Baseline
  Absolute change in low-density lipoprotein cholesterol (LDL-C) level at baseline
Low-density lipoprotein cholesterol (LDL-C) level | week 8
  Absolute change in low-density lipoprotein cholesterol (LDL-C) level at week 8
Low-density lipoprotein cholesterol (LDL-C) level | Week 26
  Absolute change in low-density lipoprotein cholesterol (LDL-C) level at week 26
Low-density lipoprotein cholesterol (LDL-C) level | Week 52
  Absolute change in low-density lipoprotein cholesterol (LDL-C) level at week 52
Low-density lipoprotein cholesterol (LDL-C) level | Baseline
  Percentage change in low-density lipoprotein cholesterol (LDL-C) level at Baseline
Low-density lipoprotein cholesterol (LDL-C) level | Week 8
  Percentage change in low-density lipoprotein cholesterol (LDL-C) level at week 8
Low-density lipoprotein cholesterol (LDL-C) level | Week 26
  Percentage change in low-density lipoprotein cholesterol (LDL-C) level at week 26
Low-density lipoprotein cholesterol (LDL-C) level | Week 52
  Percentage change in low-density lipoprotein cholesterol (LDL-C) level at week 52

SECONDARY OUTCOMES:
Rate of subject meeting LDL-C target | Week 26
  Proportion of patients meeting prespecified LDL-C goals (>50% reduction from baseline) at week 26.
Rate of subject meeting LDL-C target | Week 26
  Proportion of patients meeting prespecified LDL-C goals (<1.4mmol/l) at week 26.
Rate of subject meeting LDL-C target | Week 26
  Proportion of patients meeting prespecified LDL-C goals (<1.8mmol/L) at week 26.
12-Item Short Form Survey (SF-12) | Baseline
  Patient's quality of life as measured by SF-12 at baseline
12-Item Short Form Survey (SF-12) | Week 8
  Patient's quality of life as measured by SF-12 at week 8
12-Item Short Form Survey (SF-12) | Week 26
  Patient's quality of life as measured by SF-12 at week 26
12-Item Short Form Survey (SF-12) | Week 52
  Patient's quality of life as measured by SF-12 at week 52
Rate of major adverse cardiovascular event (MACE) | Baseline
  Occurrence of any major adverse cardiovascular event (MACE) at Baseline
Rate of major adverse cardiovascular event (MACE) | Week 8
  Occurrence of any major adverse cardiovascular event (MACE) at week 8
Rate of major adverse cardiovascular event (MACE) | Week 26
  Occurrence of any major adverse cardiovascular event (MACE) at week 26
Rate of major adverse cardiovascular event (MACE) | Week52
  Occurrence of any major adverse cardiovascular event (MACE) at week 52
Modification of lipid lowering therapy (LLT) | Week 8
  Modification of lipid lowering therapy (LLT) at week 8
Modification of lipid lowering therapy (LLT) | Week 26
  Modification of lipid lowering therapy (LLT) at week 26
Modification of lipid lowering therapy (LLT) | Week 52
  Modification of lipid lowering therapy (LLT) at week 52
Lipid Lowering Therapy adherence | Week 52
  LLT adherence, expressed in proportion of days covered, at week 52
Tolerability of Lipid Lowering Therapy | Week 52
  Rate of adverse drug event reported by subjects on lipid lowering therapy at week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Terrritories, Hong Kong

IPD SHARING:
Plan to Share IPD: No